CLINICAL TRIAL: NCT05374317
Title: An Exploratory, Pilot Study of the Safety and Immunogenicity of Reduced Doses of the US Yellow Fever Vaccine
Brief Title: Study of the Safety and Immunogenicity of Reduced Doses of the US Yellow Fever Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: FY19-26
Record Dates: First submitted 2022-03-28; First posted 2022-05-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-05

CONDITIONS: Yellow Fever Vaccination Reaction
MeSH Terms: interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard Dose (Group 1) (Active Comparator): Yellow Fever vaccine standard dose, 0.5mL.
  Interventions: Biological: Yellow Fever Vaccine
- Fractional dose (Group 2) (Experimental): Yellow Fever vaccine 1/5th standard dose, 0.1mL.
  Interventions: Biological: Yellow Fever Vaccine
- Fractional dose (Group 3) (Experimental): Yellow Fever vaccine 1/10th standard dose, 0.05mL.
  Interventions: Biological: Yellow Fever Vaccine

INTERVENTIONS:
Biological: Yellow Fever Vaccine — Administered subcutaneously once.
  Other Names: YF-VAX

SUMMARY:
This is an open-label, randomized, exploratory study to evaluate the human immune response to reduced subcutaneous (SQ) dosing of Yellow Fever vaccine compared to the standard FDA approved subcutaneous vaccination dose. The current dose of the US FDA licensed Yellow Fever vaccine is approximately 55,000 plaque-forming unit(s) (PFU) in 0.5 mL administered SQ. Using the licensed dosage as standard, investigators are evaluating reduced doses of 1/5th (0.10 mL) and 1/10th (0.05 mL) Yellow Fever vaccine (YF-VAX).

DETAILED DESCRIPTION:
Up to 150 individuals will be screened in order to randomize 90 eligible individuals to one of three groups: Group 1- YF-VAX® standard dose 0.5 mL SQ = 30 subjects; Group 2-0.10 mL (1/5th) SQ = 30 subjects; Group 3-0.05 mL (1/10th) SQ = 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females 18 to 50 years of age.
2. In good health, as determined by pertinent medical history, physical examination, vital signs, and clinical safety laboratory evaluations.
3. Female of child bearing potential: Has a negative pregnancy test and is willing to use a reliable form of contraception for the duration of the study after vaccination.
4. Negative human immunodeficiency virus (HIV) antibody screen, seronegative for hepatitis B surface antigen (HBsAg) and hepatitis C antibody (following HIV and hepatitis testing, subjects will be provided with counseling and referral for health care if any test is positive).
5. Ability to comprehend and a willingness to sign an informed consent, which includes the Health Insurance Portability and Accountability Act (HIPAA) Authorization, and a separate consent form for HIV testing.
6. Be willing to comply with all follow-up visits, testing, adverse event (AE) reporting, and completion of diary card.

Exclusion Criteria:

1. Receipt of any other investigational vaccine or investigational drug within 28 days prior to or after vaccination with YF-VAX® vaccine.
2. Have had any known flavivirus disease or receipt of any flavivirus vaccine, licensed or investigational at any time; in addition to any yellow fever vaccine, these include; Japanese Encephalitis (JE), St. Louis Encephalitis, Tick Borne Encephalitis (TBE), West Nile, Dengue, Zika virus
3. Anticipates receipt of any other vaccine within 28 days of YF-VAX®. Influenza vaccination will be permitted but not within 14 days of YF-VAX®.
4. Acute or chronic medical conditions, or medications that, in the Principal Investigator's (PI) opinion, would impair the subject's ability to respond to vaccination.
5. Hypersensitivity to any vaccine, eggs or egg products, or allergy to any component of the YF-VAX® (sorbitol, gelatin) or latex.
6. Corticosteroids even ≥20 mg/day of prednisone for ≥ 2 weeks suppresses the immune system. Low-dose corticosteroid topical products and nasal sprays used sporadically (i.e. prn--according to circumstances) are permissible.
7. History of immunosuppression, by any cause--primary or acquired immunodeficiencies, transplantation, malignant neoplasm, lymphoma, leukemia, thymoma, myasthenia gravis, radiation, immunosuppressive drugs, including antimetabolites, tumor necrosis factor (TNF)-alpha inhibitors (etanercept), interleukin-1 (IL-1) blocking agents and other monoclonal antibodies targeting immune cells (e.g., rituximab, alemtuzumab, etc), etc.
8. Receipt of or anticipates receipt of/or donation of blood or blood products for 2 months after receipt of YF-VAX®. (Note: Blood banks require a minimum 2 week interval between the receipt of this FDA licensed vaccine and blood donations; however because of the blood collections in this study, an interval of 2 months is requested).
9. Female: Pregnant (or planning to become pregnant) or breastfeeding for the duration of the study after receipt of YF-VAX®.
10. Clinically significant abnormal laboratory tests (generally 2 times the upper limit of normal or as determined by the PI).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to one year following vaccination.
  Incidence of Adverse Events of fractional doses vs standard dose of YF-VAX as determined by subject diary and clinical history and physical examination. The incidence of solicited and unsolicited adverse events will be analyzed.
Neutralizing Antibody Response | Up to one year following vaccination.
  Compare the neutralizing antibody response rate and mean of each ARM as determined by PRNT obtained at several time points. Fractional doses will be compared to the standard dose of YF-VAX. The primary data point is post vaccination day 28.

SECONDARY OUTCOMES:
Viremia | First 14 days following vaccination.
  Compare the incidence and level of viremia and mean viral load by RT-PCR (copies/mL) of fractional doses vs standard dose.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip R Pittman, M.D., M.P.H., Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- United States Army Medical Research Institute of Infectious Diseases, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monath TP, Woodall JP, Gubler DJ, Yuill TM, Mackenzie JS, Martins RM, Reiter P, Heymann DL. Yellow fever vaccine supply: a possible solution. Lancet. 2016 Apr 16;387(10028):1599-600. doi: 10.1016/S0140-6736(16)30195-7. Epub 2016 Apr 14. No abstract available. PMID 27116054
- [Background] Calisher CH, Woodall JP. Yellow Fever-More a Policy and Planning Problem than a Biological One. Emerg Infect Dis. 2016 Oct;22(10):1859-60. doi: 10.3201/eid2210.160875. Epub 2016 Oct 15. No abstract available. PMID 27479749
- [Background] Elachola H, Ditekemena J, Zhuo J, Gozzer E, Marchesini P, Rahman M, Sow S, Kattan RF, Memish ZA. Yellow fever outbreaks, vaccine shortages and the Hajj and Olympics: call for global vigilance. Lancet. 2016 Sep 17;388(10050):1155. doi: 10.1016/S0140-6736(16)31546-X. Epub 2016 Sep 5. No abstract available. PMID 27609407
- [Background] Roukens AH, Vossen AC, Bredenbeek PJ, van Dissel JT, Visser LG. Intradermally administered yellow fever vaccine at reduced dose induces a protective immune response: a randomized controlled non-inferiority trial. PLoS One. 2008 Apr 23;3(4):e1993. doi: 10.1371/journal.pone.0001993. PMID 18431480
- [Background] Slifka MK, Leung DY, Hammarlund E, Raue HP, Simpson EL, Tofte S, Baig-Lewis S, David G, Lynn H, Woolson R, Hata T, Milgrom H, Hanifin J. Transcutaneous yellow fever vaccination of subjects with or without atopic dermatitis. J Allergy Clin Immunol. 2014 Feb;133(2):439-47. doi: 10.1016/j.jaci.2013.10.037. Epub 2013 Dec 10. PMID 24331381
- [Background] Campi-Azevedo AC, de Almeida Estevam P, Coelho-Dos-Reis JG, Peruhype-Magalhaes V, Villela-Rezende G, Quaresma PF, Maia Mde L, Farias RH, Camacho LA, Freire Mda S, Galler R, Yamamura AM, Almeida LF, Lima SM, Nogueira RM, Silva Sa GR, Hokama DA, de Carvalho R, Freire RA, Filho EP, Leal Mda L, Homma A, Teixeira-Carvalho A, Martins RM, Martins-Filho OA. Subdoses of 17DD yellow fever vaccine elicit equivalent virological/immunological kinetics timeline. BMC Infect Dis. 2014 Jul 15;14:391. doi: 10.1186/1471-2334-14-391. PMID 25022840
- [Background] Wu JT, Peak CM, Leung GM, Lipsitch M. Fractional dosing of yellow fever vaccine to extend supply: a modelling study. Lancet. 2016 Dec 10;388(10062):2904-2911. doi: 10.1016/S0140-6736(16)31838-4. Epub 2016 Nov 10. PMID 27837923
- [Background] Visser LG, Roukens AH. Modelling a way out of yellow fever. Lancet. 2016 Dec 10;388(10062):2847-2848. doi: 10.1016/S0140-6736(16)31330-7. Epub 2016 Nov 10. No abstract available. PMID 27837922
- [Background] Casey RM, Harris JB, Ahuka-Mundeke S, Dixon MG, Kizito GM, Nsele PM, Umutesi G, Laven J, Kosoy O, Paluku G, Gueye AS, Hyde TB, Ewetola R, Sheria GKM, Muyembe-Tamfum JJ, Staples JE. Immunogenicity of Fractional-Dose Vaccine during a Yellow Fever Outbreak - Final Report. N Engl J Med. 2019 Aug 1;381(5):444-454. doi: 10.1056/NEJMoa1710430. Epub 2018 Feb 14. PMID 29443626
- [Background] Martins RM, Maia Mde L, Farias RH, Camacho LA, Freire MS, Galler R, Yamamura AM, Almeida LF, Lima SM, Nogueira RM, Sa GR, Hokama DA, de Carvalho R, Freire RA, Pereira Filho E, Leal Mda L, Homma A. 17DD yellow fever vaccine: a double blind, randomized clinical trial of immunogenicity and safety on a dose-response study. Hum Vaccin Immunother. 2013 Apr;9(4):879-88. doi: 10.4161/hv.22982. Epub 2013 Jan 30. PMID 23364472
- [Background] Yellow fever vaccine: WHO position on the use of fractional doses - June 2017. Wkly Epidemiol Rec. 2017 Jun 23;92(25):345-50. No abstract available. English, French. PMID 28643507
- [Background] Roukens AHE, Visser LG. Fractional-dose yellow fever vaccination: an expert review. J Travel Med. 2019 Sep 2;26(6):taz024. doi: 10.1093/jtm/taz024. PMID 30937437
- [Background] Hepburn MJ, Kortepeter MG, Pittman PR, Boudreau EF, Mangiafico JA, Buck PA, Norris SL, Anderson EL. Neutralizing antibody response to booster vaccination with the 17d yellow fever vaccine. Vaccine. 2006 Apr 5;24(15):2843-9. doi: 10.1016/j.vaccine.2005.12.055. Epub 2006 Jan 18. PMID 16494976
- [Result] Vasconcelos PF, Monath TP. Yellow Fever Remains a Potential Threat to Public Health. Vector Borne Zoonotic Dis. 2016 Aug;16(8):566-7. doi: 10.1089/vbz.2016.2031. Epub 2016 Jul 11. PMID 27400066
- See also: Addressing a Yellow Fever Vaccine Shortage — http://dx.doi.org/10.15585/mmwr.mm6617e2

DOCUMENTS (1):
  • Informed Consent Form (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT05374317/ICF_000.pdf